CLINICAL TRIAL: NCT01498393
Title: A Randomized, Placebo-Controlled Study of the 1320 nm Nd:YAG Laser for Improving the Appearance of Onychomycosis
Brief Title: 1320 nm Nd:YAG Laser for Improving the Appearance of Onychomycosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Kristen Kelly, M.D., Professor Departments of Dermatology and Surgery, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20118536
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Fungal Nail Infection
Keywords: fungal nail
MeSH Terms: conditions — Onychomycosis | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laser treatment (Other): Laser treatment to Improve the Appearance of Onychomycosis
  Interventions: Device: Laser treatment

INTERVENTIONS:
Device: Laser treatment — Laser treatment to Improve the Appearance of Onychomycosis

SUMMARY:
The purpose of this clinical study is to improve the appearance of onychomycosis and morphology of the nail (fungal infection). The researcher can use a light based therapy to gently heat the toenail infected with fungus to improve the appearance of onychomycosis.

DETAILED DESCRIPTION:
Toenail fungus (onychomycosis) is a common fungal infection of the nail that affects roughly 10% of Americans. Onychomycosis may be a precursor to many complications like ulcers, or skin infections, which may rarely result in amputation. Current treatment options have relatively limited long-term success and recurrence is common.

The researcher can determine that the laser therapy can heat the nail and destroy and decrease the fungus infecting the nail to improving the appearance of the nail.

ELIGIBILITY:
Inclusion Criteria:

* Adult Male/ female has been diagnose with fungal nail infection on both great toenails.

Exclusion Criteria:

* Any other toenail disease including, but not limited to psoriasis, lichen planus, pachyonychia congenita, etc. as determined by the investigator.
* Excessively thick or hypertrophic nails.
* Subjects with diabetes.
* Subjects that are pregnant
* Receipt of any topical therapy for onychomycosis (i.e. antifungal) within 2 weeks of enrollment, systemic therapy for onychomycosis (i.e. antifungal) within 3 months of enrollment, or any other procedures done on the test area within 6 months of enrollment.
* Subjects with impaired immune systems including, but not limited to HIV, transplant patients on immunosuppression, etc.
* Current or history of psychiatric disease that would interfere with ability to comply with the study protocol or give informed consent.
* History of alcohol or drug abuse that would interfere with ability to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improving the Appearance of fungal nail | 6 months
  Laser treatment to Improve the Appearance of Onychomycosis

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Kelly, MD, Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- Beckman Laser Institute, Irvine, California, United States

REFERENCES:
- [Result] Ortiz AE, Truong S, Serowka K, Kelly KM. A 1,320-nm Nd: YAG laser for improving the appearance of onychomycosis. Dermatol Surg. 2014 Dec;40(12):1356-60. doi: 10.1097/DSS.0000000000000189. PMID 25357174
- See also: A 1,320-nm Nd: YAG laser for improving the appearance of onychomycosis — http://www.ncbi.nlm.nih.gov/pubmed/?term=kristen+kelly